CLINICAL TRIAL: NCT03819478
Title: Effect of Protein Supplementation During Weight Loss on Older Adult Bone Health
Brief Title: Utilizing Protein During Weight Loss to Impact Physical Function and Bone
Acronym: UPLIFT-Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00038668-A; IRB00038668 (Other: Wake Forest University IRB); K25AG058804 (NIH)
Record Dates: First submitted 2019-01-18; First posted 2019-01-28 (Actual); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2021-12

CONDITIONS: Obesity; Weight Loss; Diet Modification; Aging; Weight Change, Body; Dietary Habits; Osteopenia, Osteoporosis; Bone Loss; Fractures, Bone
MeSH Terms: conditions — Obesity; Weight Loss; Body Weight Changes; Feeding Behavior; Bone Diseases, Metabolic; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: All participants will undergo a 6-month weight loss intervention of caloric restriction and supervised exercise followed by 12 months of follow-up with randomization to one of three groups (n=75/group): 1) Lower protein / higher CHO diet for the 6-month weight loss phase only (RecProt); 2) Higher protein / lower CHO diet for the 6-month weight loss phase only (6-mo HiProt); or 3) Higher protein / lower CHO diet for the 6-month weight loss and 12-month follow-up phases (18-mo HiProt).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RecProt (Active Comparator): Subjects receiving the following interventions in the parent trial (UPLIFT; NCT03074643): Lower protein / higher CHO diet for the 6-month weight loss phase. Exercise intervention months 0-6. Weight loss intervention months 0-6. Carbohydrate supplement for months 0-6 (blinded). Follow-up months 7-18.
  Interventions: Behavioral: Weight loss intervention months 0-6; Behavioral: Exercise intervention months 0-6; Dietary Supplement: NutraBio™ CarboMax Supplement
- 6-mo HiProt (Active Comparator): Subjects receiving the following interventions in the parent trial (UPLIFT; NCT03074643): Higher protein / lower CHO diet for the 6-month weight loss phase. Exercise intervention months 0-6. Weight loss intervention months 0-6. Protein supplement for months 0-6 (blinded). Follow-up months 7-18.
  Interventions: Behavioral: Weight loss intervention months 0-6; Behavioral: Exercise intervention months 0-6; Dietary Supplement: 6-month NutraBio™ 100% Whey Protein Isolate Supplement
- 18-mo HiProt (Active Comparator): Subjects receiving the following interventions in the parent trial (UPLIFT; NCT03074643):
  Higher protein / lower CHO diet for the 6-month weight loss and 12-month follow-up phases. Exercise intervention months 0-6. Weight loss intervention months 0-6. Protein supplement for months 0-6 (blinded). Protein supplement for follow-up months 7-18.
  Interventions: Behavioral: Weight loss intervention months 0-6; Behavioral: Exercise intervention months 0-6; Dietary Supplement: 18-month NutraBio™ 100% Whey Protein Isolate Supplement

INTERVENTIONS:
Behavioral: Weight loss intervention months 0-6 — All participants will undergo a dietary weight loss intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass. The weight loss intervention will incorporate nutrition education (via group and individual meetings with the study dietitian), self-monitoring skills, cognitive-behavioral strategies for promoting lifestyle behavior modifications, and planned meals. Behavioral and educational group and individual sessions will be held weekly in a 3:1 ratio (3 group and 1 individual session per month).
Behavioral: Exercise intervention months 0-6 — All participants will be expected to participate in a supervised, center-based exercise program involving moderate-intensity aerobic exercise (e.g., treadmill walking) 3 days/wk during the 6-month weight loss intervention in accordance with the American Heart Association and the American College of Sports Medicine physical activity recommendations for older adults.
Dietary Supplement: NutraBio™ CarboMax Supplement — Participants in the lower protein / higher CHO diet group (RecProt) will be provided a carbohydrate supplement (NutraBio™ CarboMax, ~50 g of carbohydrate and 220 calories) to consume daily during the 6 month weight loss intervention.
  Arms: RecProt
Dietary Supplement: 6-month NutraBio™ 100% Whey Protein Isolate Supplement — Participants in the 6-month higher protein / lower CHO diet group (6-mo HiProt) will be provided a protein supplement (NutraBio™ 100% Whey Protein Isolate, ~50 g of protein and 220 calories) to consume daily during the 6 month weight loss intervention.
  Arms: 6-mo HiProt
Dietary Supplement: 18-month NutraBio™ 100% Whey Protein Isolate Supplement — Participants in the 18-month higher protein / lower CHO diet (18-mo HiProt) will be provided a protein supplement (NutraBio™ 100% Whey Protein Isolate, ~50 g of protein and 220 calories) to consume daily during the 6 month weight loss intervention and the 12-month follow-up.
  Arms: 18-mo HiProt

SUMMARY:
This study is an ancillary study to the Utilizing Protein During Weight Loss to Impact Physical Function (UPLIFT) trial (NCT03074643) to evaluate the effects of diet composition (i.e., amount of protein and carbohydrate) during a 6-month weight loss intervention and 12-months of follow-up on bone phenotypes in obese older adults. Participants will receive either a protein or carbohydrate supplement along with a behavioral weight loss intervention.

DETAILED DESCRIPTION:
The ancillary study to the UPLIFT trial (NCT03074643) will use a 3-group design in 225 obese (body mass index [BMI] 30-45 kg/m2 or 27-<30 kg/m2 with an obesity-related risk factor), older (65-85 years) men and women at risk for disability (Short Physical Performance Battery, SPPB ≤10) who will undergo a 6-month weight loss intervention followed by a 12-month follow-up phase to test the overall hypothesis that a higher protein (1.2 g/kg body weight/day) / lower carbohydrate (CHO) diet during a 6-month weight loss intervention improves bone phenotypes compared with an isocaloric lower protein (the current Recommended Dietary Allowance (RDA), 0.8 g/kg body wt/d) / higher CHO diet, and whether continuing a higher protein / lower CHO diet for 12-months following weight loss will result in better maintenance of bone. All participants will undergo a 6-month weight loss intervention involving caloric restriction and supervised exercise followed by 12 months of follow-up with randomization to one of three groups (n=75/group): 1) Lower protein / higher CHO diet for the 6-month weight loss phase only (RecProt); 2) Higher protein / lower CHO diet for the 6-month weight loss phase only (6-mo HiProt); or 3) Higher protein / lower CHO diet for the 6-month weight loss and 12-month follow-up phases (18-mo HiProt). Vertebral and femoral volumetric bone mineral density and cortical thickness (Primary Aim) and bone marrow adipose tissue (Secondary Aim 1) will be assessed with computed tomography at baseline, 6-, and 18-months. Bone strength and fracture risk (Secondary Aim 2) will be assessed by finite element modeling at baseline, 6-, and 18-months.

ELIGIBILITY:
Subjects are recruited using inclusion and exclusion criteria of the parent trial (UPLIFT; NCT03074643).

Inclusion Criteria:

* 65-85 years
* BMI: 30-45 kg/m2 or BMI 27.0 - <30.0 AND at least one of the following risk factors:

  1. elevated waist circumference (>35 inches in women, >40 inches in men)
  2. diabetes,
  3. hypertension,
  4. dyslipidemia,
  5. or other obesity-related comorbidities: clinically manifest coronary artery disease [e.g., history of myocardial infarction, angina pectoris, coronary artery surgery, coronary artery procedures (e.g., angioplasty) if not within the past year], other atherosclerotic disease [e.g., peripheral arterial disease, abdominal aortic aneurysm, symptomatic carotid artery disease if not within the past year], sleep apnea, or osteoarthritis of the knee or hip.
* No regular resistance training and/or aerobic exercise (>20 mins/d) for past 6 months
* SPPB ≥3 to ≤10
* No contraindications for safe and optimal participation in exercise training
* Approved for participation by Medical Director (Dr. Lyles)
* Willing to provide informed consent
* Agree to all study procedures and assessments
* Willing to consume protein/CHO supplements for up to 18 months
* Able to provide own transportation to study visits and intervention sessions

Exclusion Criteria:

* Weight loss (≥5%) in past 6 months
* Dependent on cane or walker
* Cognitive impairment (Montreal Cognitive Assessment, MoCA score <22)
* Severe arthritis, or other musculoskeletal disorder
* Joint replacement or other orthopedic surgery in past year
* Uncontrolled resting hypertension (>160/90 mmHg);
* Uncontrolled diabetes (hemoglobin A1c, HbA1c ≥8.0%)
* Current or recent past (within 1 year) severe symptomatic heart disease, uncontrolled angina, stroke, chronic respiratory disease requiring oxygen; uncontrolled endocrine/metabolic disease; neurological or hematological disease; cancer requiring treatment in past year, except non-melanoma skin cancers; liver or renal disease; or clinically evident edema
* Unstable Severe Depression
* Serious conduction disorder, uncontrolled arrhythmia, or new Q waves or ST-segment depressions (>3 mm at rest or ≥2 mm with exercise)
* Abnormal kidney function (estimated glomerular rate <30 based on serum creatinine, age, gender, and race)
* Anemia (Hb<13 g/dL in men; <12 g/dL in women)
* Drug abuse or excessive alcohol use (>7 drinks/week women; >14 drinks/week men)
* Use of any tobacco or nicotine products in the past year
* Osteoporosis (T-score < -2.5 on hip or spine scan)
* Regular use of growth/steroid hormones, sex steroids or corticosteroids
* Osteoporosis medication
* Protein supplements (and unwilling to stop using for duration of study)
* Weight loss medications or procedures
* Current participation in another intervention study

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 187 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Weaver, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Geriatric Research Center at Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- RecProt: Subjects receiving the following interventions in the parent trial (NCT03074643): Lower protein / higher CHO diet for the 6-month weight loss phase. Exercise intervention months 0-6. Weight loss intervention months 0-6. Carbohydrate supplement for months 0-6 (blinded). Follow-up months 7-18.
  Weight loss intervention months 0-6: All participants underwent a dietary weight loss intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass. Weight loss intervention incorporated nutrition education (via group and individual meetings with the study dietitian), self-monitoring skills, cognitive-behavioral strategies for promoting lifestyle behavior modifications, and planned meals. Behavioral and educational group and individual sessions held weekly in a 3:1 ratio (3 group: 1 individual session/month).
  Exercise intervention months 0-6: All participants participate in a supervised, center-based exercise program involving moderate-intensity aerobic exercise (treadmill walking) 3 d/wk during the 6-month weight loss intervention in accordance with the American Heart Association and American College of Sports Medicine physical activity recommendations for older adults.
  NutraBio™ CarboMax Supplement: Participants in the RecProt group were provided a carbohydrate supplement (NutraBio™ CarboMax, ~50 g of carbohydrate, 220 calories) to consume daily during the 6 month weight loss intervention.
- 6-mo HiProt: Subjects receiving the following interventions in the parent trial (NCT03074643): Higher protein / lower CHO diet for the 6-month weight loss phase. Exercise intervention months 0-6. Weight loss intervention months 0-6. Protein supplement for months 0-6 (blinded). Follow-up months 7-18.
  Weight loss intervention months 0-6: All participants underwent a dietary weight loss intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass. Weight loss intervention incorporated nutrition education (via group and individual meetings with the study dietitian), self-monitoring skills, cognitive-behavioral strategies for promoting lifestyle behavior modifications, and planned meals. Behavioral and educational group and individual sessions held weekly in a 3:1 ratio (3 group: 1 individual session/month).
  Exercise intervention months 0-6: All participants participate in a supervised, center-based exercise program involving moderate-intensity aerobic exercise (treadmill walking) 3 d/wk during the 6-month weight loss intervention in accordance with the American Heart Association and American College of Sports Medicine physical activity recommendations for older adults.
  6-month NutraBio™ 100% Whey Protein Isolate Supplement: 6-mo HiProt participants provided a protein supplement (NutraBio™ 100% Whey Protein Isolate, 50 g of protein, 220 calories) to consume daily during the 6 month weight loss intervention.
- 18-mo HiProt: Subjects received these interventions in the parent trial (NCT03074643): Higher protein / lower CHO diet for the 6-month weight loss and 12-month follow-up. Exercise intervention months 0-6. Weight loss intervention months 0-6. Protein supplement for months 0-6 (blinded). Protein supplement for months 7-18.
  Weight loss intervention months 0-6: All participants underwent a dietary weight loss intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass. Weight loss intervention incorporated nutrition education (via group and individual meetings with the study dietitian), self-monitoring skills, cognitive-behavioral strategies for promoting lifestyle behavior modifications, and planned meals. Behavioral and educational group and individual sessions held weekly in a 3:1 ratio (3 group: 1 individual session/month).
  Exercise intervention months 0-6: All participants participate in a supervised, center-based exercise program involving moderate-intensity aerobic exercise (treadmill walking) 3 d/wk during the 6-month weight loss intervention in accordance with the American Heart Association and American College of Sports Medicine physical activity recommendations for older adults.
  18-month NutraBio™ 100% Whey Protein Isolate Supplement: 18-mo HiProt participants provided a protein supplement (NutraBio™ 100% Whey Protein Isolate, 50 g protein, 220 calories) to consume daily for the 18 months.
Period: Overall Study
Arm/Group | RecProt | 6-mo HiProt | 18-mo HiProt
Started | 62 | 62 | 63
Completed | 51 | 50 | 52
Not Completed | 11 | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RecProt | 6-mo HiProt | 18-mo HiProt | Total
Number analyzed (Participants) | 62 | 62 | 63 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (4.4) | 71.8 (4.5) | 70.5 (3.9) | 71.0 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 42 | 124
  Male | 21 | 21 | 21 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 61 | 62 | 63 | 186
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 14 | 19 | 45
  White | 48 | 47 | 43 | 138
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.8 (4.6) | 34.3 (3.5) | 34.3 (4.2) | 34.2 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: 18-month Change From Baseline in Total Hip Trabecular Volumetric Bone Mineral Density Assessed by Computed Tomography (CT) in mg/cm^3
Description: To determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet on the 18-month change from baseline in total hip trabecular volumetric bone mineral density (vBMD). Total hip trabecular vBMD (in mg/cm^3) was measured from the baseline and 18-month quantitative CT scans using the Mindways Model 3 phantom to calibrate the vBMD measures. The 18-month change in total hip trabecular vBMD from baseline is reported for this outcome measure.
Time Frame: Change from Baseline to Month 18
Measure: Least Squares Mean (Standard Error); unit: mg/cm^3
Arm/Group | RecProt | 6-mo HiProt | 18-mo HiProt
Number analyzed (Participants) | 38 | 38 | 38
mg/cm^3 | -0.91 (1.34) | -1.77 (1.40) | -0.03 (1.44)
Statistical Analysis 1: Comparison: RecProt vs 18-mo HiProt; Test type: Superiority; p = 0.4880, ANCOVA; Adjusted for age, sex, race, and baseline bone measure
Statistical Analysis 2: Comparison: 6-mo HiProt vs 18-mo HiProt; Test type: Superiority; p = 0.1683, ANCOVA; Adjusted for age, sex, race, and baseline bone measure

2. Secondary Outcome: 6-month Change From Baseline in Percentage of Adipose Tissue Within the Lumbar Spine Bone Marrow as Assessed by Dual-energy Computed Tomography Algorithm
Description: Percentage of adipose tissue within the lumbar spine bone marrow as assessed by a dual-energy computed tomography (CT) algorithm to determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet. Percentage of adipose tissue within the bone marrow was measured from the baseline and 6-month dual-energy CT scans using a Mindways Model 3 phantom for calibration. The 6-month change in percentage of adipose tissue within the lumbar spine bone marrow from baseline is reported for this outcome measure.
Time Frame: Change from Baseline to Month 6
Population: The two protein supplement groups ("6-mo HiProt" and "18-mo HiProt") are combined into a single "HiProt" group as both groups received the same intervention for months 0-6, and this outcome measure is reporting the change from Baseline to Month 6.
Measure: Least Squares Mean (Standard Error); unit: percentage of bone marrow adiposity
Groups:
- RecProt: Subjects receiving the following interventions in the parent trial (NCT03074643): Lower protein / higher CHO diet for the 6-month weight loss phase. Exercise intervention months 0-6. Weight loss intervention months 0-6. Carbohydrate supplement for months 0-6 (blinded).
  Weight loss intervention months 0-6: All participants underwent a dietary weight loss intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass. Weight loss intervention incorporated nutrition education (via group and individual meetings with the study dietitian), self-monitoring skills, cognitive-behavioral strategies for promoting lifestyle behavior modifications, and planned meals. Behavioral and educational group and individual sessions held weekly in a 3:1 ratio (3 group: 1 individual session/month).
  Exercise intervention months 0-6: All participants participate in a supervised, center-based exercise program involving moderate-intensity aerobic exercise (treadmill walking) 3 d/wk during the 6-month weight loss intervention in accordance with the American Heart Association and American College of Sports Medicine physical activity recommendations for older adults.
  NutraBio™ CarboMax Supplement: Participants in the RecProt group were provided a carbohydrate supplement (NutraBio™ CarboMax, ~50 g of carbohydrate, 220 calories) to consume daily during the 6 month weight loss intervention.
- HiProt: Subjects receiving the following interventions in the parent trial (NCT03074643): Higher protein / lower CHO diet for the 6-month weight loss phase. Exercise intervention months 0-6. Weight loss intervention months 0-6. Protein supplement for months 0-6 (blinded).
  Weight loss intervention months 0-6: All participants underwent a dietary weight loss intervention designed to elicit behavioral changes leading to decreased caloric intake sufficient to yield a ~10% loss of initial body mass. Weight loss intervention incorporated nutrition education (via group and individual meetings with the study dietitian), self-monitoring skills, cognitive-behavioral strategies for promoting lifestyle behavior modifications, and planned meals. Behavioral and educational group and individual sessions held weekly in a 3:1 ratio (3 group: 1 individual session/month).
  Exercise intervention months 0-6: All participants participate in a supervised, center-based exercise program involving moderate-intensity aerobic exercise (treadmill walking) 3 d/wk during the 6-month weight loss intervention in accordance with the American Heart Association and American College of Sports Medicine physical activity recommendations for older adults.
  6-month NutraBio™ 100% Whey Protein Isolate Supplement: 6-mo HiProt participants provided a protein supplement (NutraBio™ 100% Whey Protein Isolate, 50 g of protein, 220 calories) to consume daily during the 6 month weight loss intervention.
Arm/Group | RecProt | HiProt
Number analyzed (Participants) | 41 | 89
percentage of bone marrow adiposity | 7.42 (4.06) | 6.45 (3.81)
Statistical Analysis 1: Comparison: RecProt vs HiProt; Test type: Superiority; p = 0.7636, ANCOVA; Adjusted for age, sex, race, and baseline bone measure

3. Secondary Outcome: 18-month Change From Baseline in Percentage of Adipose Tissue Within the Lumbar Spine Bone Marrow as Assessed by Dual-energy Computed Tomography Algorithm
Description: Percentage of adipose tissue within the lumbar spine bone marrow as assessed by a dual-energy computed tomography (CT) algorithm to determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet. Percentage of adipose tissue within the bone marrow was measured from the baseline and 18-month dual-energy CT scans using a Mindways Model 3 phantom for calibration. The 18-month change in percentage of adipose tissue within the lumbar spine bone marrow from baseline is reported for this outcome measure.
Time Frame: Change from Baseline to Month 18
Measure: Least Squares Mean (Standard Error); unit: percentage of bone marrow adiposity
Arm/Group | RecProt | 6-mo HiProt | 18-mo HiProt
Number analyzed (Participants) | 36 | 39 | 38
percentage of bone marrow adiposity | -0.20 (3.69) | -9.96 (3.80) | -5.17 (3.93)
Statistical Analysis 1: Comparison: RecProt vs 18-mo HiProt; Test type: Superiority; p = 0.1584, ANCOVA; Adjusted for age, sex, race, and baseline bone measure
Statistical Analysis 2: Comparison: 6-mo HiProt vs 18-mo HiProt; Test type: Superiority; p = 0.1623, ANCOVA; Adjusted for age, sex, race, and baseline bone measure

4. Secondary Outcome: 6-month Change From Baseline in Femoral Bone Strength in kN
Description: Subject-specific finite element models were created from the baseline and 6-month CT scans and femoral bone strength was assessed from a simulated test of a sideways fall. Bone strength was measured as the peak section force extracted at the femoral neck to determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet on the 6-month change from baseline in femoral bone strength.
Time Frame: Change from Baseline to Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kN
Arm/Group | RecProt | HiProt
Number analyzed (Participants) | 42 | 87
kN | -0.02 (0.08) | 0.10 (0.07)
Statistical Analysis 1: Comparison: RecProt vs HiProt; Test type: Superiority; p = 0.0350, ANCOVA; Adjusted for age, sex, race, and baseline bone measure

5. Secondary Outcome: 18-month Change From Baseline in Femoral Bone Strength in kN
Description: Subject-specific finite element models were created from the baseline and 18-month CT scans and femoral bone strength was assessed from a simulated test of a sideways fall. Bone strength was measured as the peak section force extracted at the femoral neck to determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet on the 18-month change from baseline in femoral bone strength.
Time Frame: Change from Baseline to Month 18
Measure: Least Squares Mean (Standard Error); unit: kN
Arm/Group | RecProt | 6-mo HiProt | 18-mo HiProt
Number analyzed (Participants) | 38 | 38 | 38
kN | -0.02 (0.10) | 0.03 (0.11) | 0.09 (0.11)
Statistical Analysis 1: Comparison: RecProt vs 18-mo HiProt; Test type: Superiority; p = 0.2422, ANCOVA; Adjusted for age, sex, race, and baseline bone measure
Statistical Analysis 2: Comparison: 6-mo HiProt vs 18-mo HiProt; Test type: Superiority; p = 0.5082, ANCOVA; Adjusted for age, sex, race, and baseline bone measure

6. Secondary Outcome: 18-month Change From Baseline in Femoral Cortical Thickness Assessed by Computed Tomography (CT) in mm
Description: Cortical thickness of the proximal femur was assessed by a computed tomography (CT) based algorithm to determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet on the 18-month change from baseline in femoral cortical thickness. Cortical thickness was measured from the baseline and 18-month CT scans, and the 18-month change from baseline (in mm) is reported for this outcome measure.
Time Frame: Change from Baseline to Month 18
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | RecProt | 6-mo HiProt | 18-mo HiProt
Number analyzed (Participants) | 41 | 42 | 42
mm | 0.02 (0.02) | 0.02 (0.02) | 0.01 (0.03)
Statistical Analysis 1: Comparison: RecProt vs 18-mo HiProt; Test type: Superiority; p = 0.5119, ANCOVA; Adjusted for age, sex, race, and baseline bone measure
Statistical Analysis 2: Comparison: 6-mo HiProt vs 18-mo HiProt; Test type: Superiority; p = 0.4902, ANCOVA; Adjusted for age, sex, race, and baseline bone measure

7. Secondary Outcome: 6-month Change From Baseline in Femoral Cortical Thickness Assessed by Computed Tomography (CT) in mm
Description: Cortical thickness of the proximal femur was assessed by a computed tomography (CT) based algorithm to determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet on the 6-month change from baseline in femoral cortical thickness. Cortical thickness was measured from the baseline and 6-month CT scans, and the 6-month change from baseline (in mm) is reported for this outcome measure.
Time Frame: Change from Baseline to Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | RecProt | HiProt
Number analyzed (Participants) | 46 | 96
mm | 0.01 (0.02) | 0.01 (0.02)
Statistical Analysis 1: Comparison: RecProt vs HiProt; Test type: Superiority; p = 0.8500, ANCOVA; Adjusted for age, sex, race, and baseline bone measure

8. Secondary Outcome: 18-month Change From Baseline in Vertebral Volumetric Bone Mineral Density in the Lumbar Spine Assessed by Computed Tomography (CT) in mg/cm^3
Description: To determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet on the 18-month change from baseline in vertebral volumetric bone mineral density (vBMD) in the lumbar spine. Trabecular vBMD (in mg/cm^3) was measured from the baseline and 18-month quantitative CT scans using the Mindways Model 3 phantom to calibrate the vertebral vBMD measures. The 18-month change in vertebral vBMD in the lumbar spine from baseline is reported for this outcome measure.
Time Frame: Change from Baseline to Month 18
Measure: Least Squares Mean (Standard Error); unit: mg/cm^3
Arm/Group | RecProt | 6-mo HiProt | 18-mo HiProt
Number analyzed (Participants) | 42 | 44 | 48
mg/cm^3 | -1.40 (1.48) | -0.39 (1.54) | -2.59 (1.57)
Statistical Analysis 1: Comparison: RecProt vs 18-mo HiProt; Test type: Superiority; p = 0.3685, ANCOVA; Adjusted for age, sex, race, and baseline bone measure
Statistical Analysis 2: Comparison: 6-mo HiProt vs 18-mo HiProt; Test type: Superiority; p = 0.0894, ANCOVA; Adjusted for age, sex, race, and baseline bone measure

9. Secondary Outcome: 6-month Change From Baseline in Vertebral Volumetric Bone Mineral Density in the Lumbar Spine Assessed by Computed Tomography (CT) in mg/cm^3
Description: To determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet on the 6-month change from baseline in vertebral volumetric bone mineral density (vBMD) in the lumbar spine. Trabecular vBMD (in mg/cm^3) was measured from the baseline and 6-month quantitative CT scans using the Mindways Model 3 phantom to calibrate the vertebral vBMD measures. The 6-month change in vertebral vBMD in the lumbar spine from baseline is reported for this outcome measure.
Time Frame: Change from Baseline to Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/cm^3
Arm/Group | RecProt | HiProt
Number analyzed (Participants) | 49 | 108
mg/cm^3 | 2.87 (1.48) | 3.56 (1.41)
Statistical Analysis 1: Comparison: RecProt vs HiProt; Test type: Superiority; p = 0.5334, ANCOVA; Adjusted for age, sex, race, and baseline bone measure

10. Secondary Outcome: 6-month Change From Baseline in Total Hip Trabecular Volumetric Bone Mineral Density Assessed by Computed Tomography (CT) in mg/cm^3
Description: To determine the effects of a higher protein / lower CHO diet vs. lower protein / higher CHO diet on the 6-month change from baseline in total hip trabecular volumetric bone mineral density (vBMD). Total hip trabecular vBMD (in mg/cm^3) was measured from the baseline and 6-month quantitative CT scans using the Mindways Model 3 phantom to calibrate the vBMD measures. The 6-month change in total hip trabecular vBMD from baseline is reported for this outcome measure.
Time Frame: Change from Baseline to Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/cm^3
Arm/Group | RecProt | HiProt
Number analyzed (Participants) | 42 | 87
mg/cm^3 | 0.34 (1.12) | 1.59 (1.05)
Statistical Analysis 1: Comparison: RecProt vs HiProt; Test type: Superiority; p = 0.1573, ANCOVA; Adjusted for age, sex, race, and baseline bone measure

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | RecProt | 6-mo HiProt | 18-mo HiProt
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62 | 0/63
Serious Adverse Events (participants affected / at risk) | 8/62 | 5/62 | 5/63
Other Adverse Events (participants affected / at risk) | 17/62 | 14/62 | 11/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RecProt (N=62) | 6-mo HiProt (N=62) | 18-mo HiProt (N=63)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cognitive Disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Knee Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Transurethral Resection Of Prostrate (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Shoulder Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Revision of Knee Replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hip Replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Umbilical Hernia Repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Reverse Shoulder Arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RecProt (N=62) | 6-mo HiProt (N=62) | 18-mo HiProt (N=63)
Sinusitis (Infections and infestations) | 7 (8) | 2 (2) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 1 (1) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 7 (9) | 6 (6) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
We initially planned to end recruitment in August of 2020. However, our institution paused all in-person research from March 13, 2020 through May 31, 2020 due to the COVID19 pandemic. We extended our recruitment window through September 2020 but did not reach our target enrollment. The COVID19 pandemic also affected participant follow-up (a large number of out of window visits and a few who refused to return for in-person visits). The 6-month intervention also had to go remote for ~4 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT03819478/Prot_002.pdf
  • Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT03819478/SAP_003.pdf
  • Informed Consent Form (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT03819478/ICF_001.pdf